CLINICAL TRIAL: NCT00249509
Title: Marijuana Pharmacotherapies: Controlled Clinical Trials With Nefazodone and Bupropion
Brief Title: Effectiveness of Nefazodone and Bupropion in Treating Marijuana Dependent Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Frances R. Levin, M.D, NYSPI
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-13191-1; R01-DA013191-1; DPMC; R01DA013191 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2011-03

CONDITIONS: Marijuana Abuse
Keywords: marijuana dependence
MeSH Terms: conditions — Marijuana Abuse | interventions — nefazodone; Bupropion

INTERVENTIONS:
Drug: Nefazodone
Drug: Bupropion

SUMMARY:
Recent research has identified the following withdrawal symptoms to be associated with abruptly stopping marijuana use: anxiety, irritability, bodily aches and pains, and difficulty sleeping. These symptoms resemble those of both depression and nicotine withdrawal, suggesting that a similar treatment drug may be useful. This study will evaluate the effectiveness of two antidepressant drugs, bupropion and nefazodone, in reducing withdrawal symptoms in marijuana dependent individuals.

DETAILED DESCRIPTION:
There have been few controlled studies that focus on treatments for marijuana dependence. The symptoms associated with marijuana withdrawal, including anxiety, irritability, bodily aches and pains, and difficulty sleeping, resemble those caused by depression and nicotine withdrawal. Therefore, antidepressant or nicotine withdrawal medications may be effective in treating marijuana dependence. Nefazodone and bupropion are two medications currently used to treat depression. The purpose of this study is to determine the effectiveness of nefazodone and bupropion in alleviating marijuana withdrawal symptoms. In addition, this study will evaluate whether these medications successfully treat marijuana dependent individuals in terms of treatment adherence and drug abstinence.

Participants in this double-blind trial will be randomly assigned to receive nefazodone, bupropion, or placebo. Daily doses of medication will be provided to participants in dated pill boxes; pill boxes will then be returned to the study nurse at each study visit. Medication will be taken in three daily doses; one of the doses will be a nonmedicated pill. Nefazodone will initially be given at a dose of 150 mg per day, which participants will take at bedtime. Every 5 days, the daily dose will increase by 150 mg, to a maximal dose of 600 mg of nefazodone per day. Bupropion will be given at an initial dose of 150 mg, which participants will take in the morning. After 3 days, the daily dose will increase to a total dose of 300 mg of bupropion per day.

Study visits will occur daily, at which time participants will complete drug use and withdrawal symptom reports. In addition, participants will partake in weekly therapy visits, which will consist of four sessions of motivational enhancement therapy followed by sessions of relapse prevention therapy. Bi-weekly psychiatry visits will include evaluations on substance use behavior and overall clinical symptoms, and will last 15-30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for current marijuana dependence
* Uses at least 5 marijuana joints per week
* Currently seeking treatment for marijuana dependence
* Used marijuana in a maladaptive pattern in the 6 months prior to study entry

Exclusion Criteria:

* History of seizures or unexplained loss of consciousness
* Significant and unstable psychiatric condition (e.g., schizophrenia, bipolar disorder)
* Chronic organic mental disorder
* Dependent on any substances of abuse other than marijuana
* Currently at significant suicidal risk
* Unstable physical disorder that may represent a severe untreated condition, such as hypertension (blood pressure greater than 150/90), elevated transaminase levels, or unstable diabetes
* Current or suspected coronary vascular disease
* Has taken a monoamine oxidase inhibitor in the 2 weeks prior to study entry
* Currently taking terfenedine, cisapride, astemizole, or pimozide
* History of an allergic reaction to bupropion or nefazodone
* If female, pregnant, breastfeeding, or unwilling to use an adequate method of contraception for the duration of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132
Dates: Start 2000-09; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Marijuana use

SECONDARY OUTCOMES:
Marijuana withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: David Mcdowell, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- See also: Click here for more information about the Substance Treatment and Research Service — http://stars.columbia.edu/